CLINICAL TRIAL: NCT05806606
Title: The Effects and Cost-effectiveness of a Dyadic Empowerment-based Heart Failure Management Program (De-HF) on Self-care, HRQL and Hospital Readmission: A Randomized Controlled Trial
Brief Title: Effect and Cost Effectiveness of a Dyadic Empowerment-based Heart Failure Management Program for Self-care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DE-HF
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Self Care; Empowerment; Transitional Care; Disease Management
Keywords: Heart Failure; Self Care; Empowerment; Dyadic; Disease management; Transitional care
MeSH Terms: conditions — Heart Failure; Empowerment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: It is a double-blind study. A research nurse will identify potential subjects from the Clinical Management System.
  Eligible patients and their primary carers will be invited to participate during their hospital stay. After obtaining their written informed consent, the research nurse will collect their baseline demographic data and administer the following outcome measures in a face-to-face interview.
  The care dyads will be randomized by computer generated sequence in a 1:1 allocation ratio to receive either the De-HF or the HF dyadic educational program. To ensure double blinding, the dyads will not know whether they are participating in the test or control intervention, and the outcome measurement will be conducted by another research assistant without knowing the assigned group of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic Empowerment-based Heart Failure program (De-HF) (Experimental): The 16-week De-HF Program is delivered on a dyadic basis. The program consists of three core elements: i) joint dyadic interview in a home visit (1st-2nd week), ii) five ICT-enhanced empowerment-based modules (3rd-12th week; 2 sessions/ each module), and iii) post-module telephone follow-up (13th-16th week). The overall aim of the dyadic interview is to understand their usual pattern of collaboration, deficits, strengths and competing concerns in disease management. This is followed by the empowerment modules with the purpose to help the care dyads to get a consensus in disease interpretation (1st session: Perceptual and Cognitive Empowerment Session) and develop collaborative goal attainment process (2nd Session: Collaborative Gaol-Setting Process). This will be followed by two bi-weekly telephone calls to the care dyads using a speaker phone to monitor their level of goal attainment for the five modules, and to give further advice and counselling.
  Interventions: Other: Dyadic empowerment based heart failure management program
- Dyadic education program (Active Comparator): The 16-week HF education program comprises a home visit, five bi-weekly online training sessions, and the subsequent telephone follow-up for the care dyads. The nurse will first assess how they manage HF in terms of medication compliance, fluid and dietary control, symptom monitoring and responses in a home visit and clarify their major misconceptions in self-care. This will be followed by five bi-weekly online education sessions on the same topics as the empowerment modules in the De-HF program.
  Interventions: Other: Dyadic education program

INTERVENTIONS:
Other: Dyadic empowerment based heart failure management program — The 16-week De-HF Program is delivered on a dyadic basis, The program consists of three core elements: i) joint dyadic interview in a home visit (1st-2nd week), ii) five ICT-enhanced empowerment-based modules (3rd-12th week; 2 sessions/ each module), and iii) post-module telephone follow-up (13th-16th week). The overall aim of the dyadic interview is to understand their usual pattern of collaboration, deficits, strengths and competing concerns in disease management. This is followed by the empowerment modules with the purpose to help the care dyads to get a consensus in disease interpretation (1st session: Perceptual and Cognitive Empowerment Session) and develop collaborative goal attainment process (2nd Session: Collaborative Gaol-Setting Process). This will be followed by two bi-weekly telephone calls to the care dyads using a speaker phone to monitor their level of goal attainment for the five modules, and to give further advice and counselling.
  Arms: Dyadic Empowerment-based Heart Failure program (De-HF)
Other: Dyadic education program — The 16-week HF education program comprises a home visit, five bi-weekly online training sessions, and the subsequent telephone follow-up for the care dyads. The nurse will first assess how they manage HF in terms of medication compliance, fluid and dietary control, symptom monitoring and responses in a home visit and clarify their major misconceptions in self-care. This will be followed by five bi-weekly online education sessions on the same topics as the empowerment modules in the De-HF program.
  Arms: Dyadic education program

SUMMARY:
Global population aging has drastically increased healthcare spending worldwide, with the greatest portion going to hospital and community health services. Heart failure (HF), as the final form of many cardiovascular diseases resulting from insufficient myocardial pumping. Ineffective self-care is consistently identified as the major modifiable risk factor for HF decompensation requiring hospitalization. It refers to an active cognitive process that influence patients' engagement in self-care maintenance, symptom perception and self-care management. However, current studies pay much focus on interventions such as motivational interviewing and behavioural activation to enhance the HF-related self-care and health outcomes which only produces short-term benefits. In fact, the lack of a sustainable effect from the self-care supportive interventions might be related the use of patient-centric design in these studies, which totally ignores the fact that HF management takes place in a dyadic context. To advance, active strategies were adopted to mobilize collaborative effort of the dyad in actual disease management.

This study aims to evaluate the effects and cost-effectiveness of a Dyadic empowerment-based Heart Failure Management Program (De-HF) for self-care, health outcomes, and health service utilization among HF patients who require family support after hospital discharge. The De-HF program is based on the Theory of Dyadic Illness Management to enhance the congruence in illness perception and active dyadic collaboration in managing HF via both face-to-face and online platforms.

DETAILED DESCRIPTION:
This is a mixed-method RCT to evaluate the effects and cost-effectiveness of the Dyadic Empowerment Heart Failure Program on improving self-care, health-related quality of life, hospital readmission and emergency room utilization among the HF patients discharged from the hospital. The study will be conducted in three regional hospital in Hong Kong, with subjects to be recruited from the in-patient setting.

The subjects need to be aged 18 or above, with an index diagnosis of HF in admission, at New York Heart Association Classification Class II-IV, to be discharged home and with Abbreviated Mental Test score >6.

The caregiver need to the primary caregivers, co-residing with the patients, and have access to smartphone. Power analysis estimate the sample size as 232 care dyads who will be allocated in a 1:1 ratio to receive the DE-HF Program of the HF dyadic education intervention. The 16-week De-HF program will be commenced within 2 weeks of discharge. It will starts with a dyadic interview in a home visit to identify the usual pattern of collaboration, deficits, strengths and competing concerns in disease management. This is followed by five empowerment modules with the purpose to help the care dyads to get a consensus and optimize their joint efforts in disease management. The five topics include symptom management, dietary and fluid modification, medication management, symptom management, activity and exercise. For each module, there are two sessions for i) perception and cognitive empowerment and ii) develop collaborative goal attainment process. Upon the completion of the ten sessions, two bi-weekly telephone calls will be made to the care dyads to monitor their level of goal attainment, and to give further advice and counselling. The 16-week dyadic education program will cover one home visit to assess their disease management at home, and this will be followed by five standard bi-weekly online education session on the same topics as the modules in the De-HF program. Outcome evaluation will take place at baseline, post-test 16th week, 24th week and 32rd week with validated measure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Confirmed medical diagnosis of Heart Failure by a cardiologist of at least 3 months
* New York Heart Association (NYHA) Class II-IV symptoms
* Discharged home after an admission to the recruitment setting
* Carer co-residing with the patients in the same household
* Carer self-identified as the primary carer for the patients
* Both the patient and the carer having adequate cognitive ability (as indicated by an Abbreviated Test Score of >6)
* Have at least one Smartphone or device to access the online meetings and videos

Exclusion Criteria:

* Not living with primary caregiver
* With end-stage renal disease relying on hemodialysis rather than HF medications to regulate fluid volume.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure (MLHF) questionnaire | Baseline
  Measure the disease-specific HRQL (primary outcome of the HF patient), covering the physical and emotional health of HF patients. There are 21 items and each item is rated from 0 to 5, with higher scores indicating poor health.
Minnesota Living with Heart Failure (MLHF) questionnaire | 16th week
  Measure the disease-specific HRQL (primary outcome of the HF patient), covering the physical and emotional health of HF patients. There are 21 items and each item is rated from 0 to 5, with higher scores indicating poor health.
Minnesota Living with Heart Failure (MLHF) questionnaire | 24th week
  Measure the disease-specific HRQL (primary outcome of the HF patient), covering the physical and emotional health of HF patients. There are 21 items and each item is rated from 0 to 5, with higher scores indicating poor health.
Minnesota Living with Heart Failure (MLHF) questionnaire | 32nd week
  Measure the disease-specific HRQL (primary outcome of the HF patient), covering the physical and emotional health of HF patients. There are 21 items and each item is rated from 0 to 5, with higher scores indicating poor health.
The EuroQoL-5D-5L instruments | Baseline
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems, moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5D-5L instruments | 16th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems, moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5D-5L instruments | 24th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems, moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5D-5L instruments | 32nd week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems, moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.

SECONDARY OUTCOMES:
Self-Care Heart Failure Index (SCHFI, v.7.2) | Baseline
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 16th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 24th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 32nd week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Shared Care Instrument-Revised (SCI-3) | Baseline
  Measure the level of shared care in terms of communication, decision-making, and reciprocity of care dyads. Each item is rated from zero to five (completely agree, mostly agree, slightly agree, slightly disagree, mostly disagree, and completely disagree), with higher scores representing better shared care.
Shared Care Instrument-Revised (SCI-3) | 16th week
  Measure the level of shared care in terms of communication, decision-making, and reciprocity of care dyads. Each item is rated from zero to five (completely agree, mostly agree, slightly agree, slightly disagree, mostly disagree, and completely disagree), with higher scores representing better shared care.
Shared Care Instrument-Revised (SCI-3) | 24th week
  Measure the level of shared care in terms of communication, decision-making, and reciprocity of care dyads. Each item is rated from zero to five (completely agree, mostly agree, slightly agree, slightly disagree, mostly disagree, and completely disagree), with higher scores representing better shared care.
Shared Care Instrument-Revised (SCI-3) | 32nd week
  Measure the level of shared care in terms of communication, decision-making, and reciprocity of care dyads. Each item is rated from zero to five (completely agree, mostly agree, slightly agree, slightly disagree, mostly disagree, and completely disagree), with higher scores representing better shared care.
Control Attitude Scale Revised (CAS-R) | Baseline
  Measure the perceived control in disease management. Each item was rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) and summed to create a total score after two negative items were reverse coded. The possible total score ranges from 8 to 40 with a higher score indicating higher perceived controllability.
Control Attitude Scale Revised (CAS-R) | 16th week
  Measure the perceived control in disease management. Each item was rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) and summed to create a total score after two negative items were reverse coded. The possible total score ranges from 8 to 40 with a higher score indicating higher perceived controllability.
Control Attitude Scale Revised (CAS-R) | 24th week
  Measure the perceived control in disease management. Each item was rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) and summed to create a total score after two negative items were reverse coded. The possible total score ranges from 8 to 40 with a higher score indicating higher perceived controllability.
Control Attitude Scale Revised (CAS-R) | 32nd week
  Measure the perceived control in disease management. Each item was rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) and summed to create a total score after two negative items were reverse coded. The possible total score ranges from 8 to 40 with a higher score indicating higher perceived controllability.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Tseung Kwan O Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.

REFERENCES:
- [Result] Groenewegen A, Rutten FH, Mosterd A, Hoes AW. Epidemiology of heart failure. Eur J Heart Fail. 2020 Aug;22(8):1342-1356. doi: 10.1002/ejhf.1858. Epub 2020 Jun 1. PMID 32483830
- [Result] Ryan CJ, Bierle RS, Vuckovic KM. The Three Rs for Preventing Heart Failure Readmission: Review, Reassess, and Reeducate. Crit Care Nurse. 2019 Apr;39(2):85-93. doi: 10.4037/ccn2019345. PMID 30936132
- [Result] Riegel B, Barbaranelli C, Carlson B, Sethares KA, Daus M, Moser DK, Miller J, Osokpo OH, Lee S, Brown S, Vellone E. Psychometric Testing of the Revised Self-Care of Heart Failure Index. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):183-192. doi: 10.1097/JCN.0000000000000543. PMID 30303894
- [Result] Jonkman NH, Westland H, Groenwold RH, Agren S, Atienza F, Blue L, Bruggink-Andre de la Porte PW, DeWalt DA, Hebert PL, Heisler M, Jaarsma T, Kempen GI, Leventhal ME, Lok DJ, Martensson J, Muniz J, Otsu H, Peters-Klimm F, Rich MW, Riegel B, Stromberg A, Tsuyuki RT, van Veldhuisen DJ, Trappenburg JC, Schuurmans MJ, Hoes AW. Do Self-Management Interventions Work in Patients With Heart Failure? An Individual Patient Data Meta-Analysis. Circulation. 2016 Mar 22;133(12):1189-98. doi: 10.1161/CIRCULATIONAHA.115.018006. Epub 2016 Feb 12. PMID 26873943
- [Result] Buck HG, Harkness K, Wion R, Carroll SL, Cosman T, Kaasalainen S, Kryworuchko J, McGillion M, O'Keefe-McCarthy S, Sherifali D, Strachan PH, Arthur HM. Caregivers' contributions to heart failure self-care: a systematic review. Eur J Cardiovasc Nurs. 2015 Feb;14(1):79-89. doi: 10.1177/1474515113518434. Epub 2014 Jan 6. PMID 24399843
- [Result] Strachan PH, Currie K, Harkness K, Spaling M, Clark AM. Context matters in heart failure self-care: a qualitative systematic review. J Card Fail. 2014 Jun;20(6):448-55. doi: 10.1016/j.cardfail.2014.03.010. Epub 2014 Apr 13. PMID 24735549
- [Result] Clark AM, Spaling M, Harkness K, Spiers J, Strachan PH, Thompson DR, Currie K. Determinants of effective heart failure self-care: a systematic review of patients' and caregivers' perceptions. Heart. 2014 May;100(9):716-21. doi: 10.1136/heartjnl-2013-304852. Epub 2014 Feb 18. PMID 24548920
- [Result] Buck HG, Stromberg A, Chung ML, Donovan KA, Harkness K, Howard AM, Kato N, Polo R, Evangelista LS. A systematic review of heart failure dyadic self-care interventions focusing on intervention components, contexts, and outcomes. Int J Nurs Stud. 2018 Jan;77:232-242. doi: 10.1016/j.ijnurstu.2017.10.007. Epub 2017 Oct 19. PMID 29128777
- [Result] Vellone E, Rebora P, Ausili D, Zeffiro V, Pucciarelli G, Caggianelli G, Masci S, Alvaro R, Riegel B. Motivational interviewing to improve self-care in heart failure patients (MOTIVATE-HF): a randomized controlled trial. ESC Heart Fail. 2020 Jun;7(3):1309-1318. doi: 10.1002/ehf2.12733. Epub 2020 Apr 28. PMID 32343483
- [Result] Lyons KS, Lee CS. The Theory of Dyadic Illness Management. J Fam Nurs. 2018 Feb;24(1):8-28. doi: 10.1177/1074840717745669. Epub 2018 Jan 20. PMID 29353528
- [Result] Sebern M, Riegel B. Contributions of supportive relationships to heart failure self-care. Eur J Cardiovasc Nurs. 2009 Jun;8(2):97-104. doi: 10.1016/j.ejcnurse.2008.07.004. Epub 2008 Aug 15. PMID 18706865
- [Result] Srisuk N, Cameron J, Ski CF, Thompson DR. Randomized controlled trial of family-based education for patients with heart failure and their carers. J Adv Nurs. 2017 Apr;73(4):857-870. doi: 10.1111/jan.13192. Epub 2016 Nov 30. PMID 27779768
- [Result] Sebern MD, Woda A. Shared care dyadic intervention: outcome patterns for heart failure care partners. West J Nurs Res. 2012 Apr;34(3):289-316. doi: 10.1177/0193945911399088. Epub 2011 Mar 7. PMID 21383082
- [Result] Boczor S, Daubmann A, Eisele M, Blozik E, Scherer M. Quality of life assessment in patients with heart failure: validity of the German version of the generic EQ-5D-5L. BMC Public Health. 2019 Nov 6;19(1):1464. doi: 10.1186/s12889-019-7623-2. PMID 31694584
- [Result] Tidermark J, Bergstrom G, Svensson O, Tornkvist H, Ponzer S. Responsiveness of the EuroQol (EQ 5-D) and the SF-36 in elderly patients with displaced femoral neck fractures. Qual Life Res. 2003 Dec;12(8):1069-79. doi: 10.1023/a:1026193812514. PMID 14651424
- [Result] Yu DS, Lee DT, Stewart S, Thompson DR, Choi KC, Yu CM. Effect of Nurse-Implemented Transitional Care for Chinese Individuals with Chronic Heart Failure in Hong Kong: A Randomized Controlled Trial. J Am Geriatr Soc. 2015 Aug;63(8):1583-93. doi: 10.1111/jgs.13533. PMID 26289684
- [Result] Yu DS, Li PW, Zhang F, Cheng ST, Ng TK, Judge KS. The effects of a dyadic strength-based empowerment program on the health outcomes of people with mild cognitive impairment and their family caregivers: a randomized controlled trial. Clin Interv Aging. 2019 Oct 4;14:1705-1717. doi: 10.2147/CIA.S213006. eCollection 2019. PMID 31686796
- [Result] Jaarsma T, Hill L, Bayes-Genis A, La Rocca HB, Castiello T, Celutkiene J, Marques-Sule E, Plymen CM, Piper SE, Riegel B, Rutten FH, Ben Gal T, Bauersachs J, Coats AJS, Chioncel O, Lopatin Y, Lund LH, Lainscak M, Moura B, Mullens W, Piepoli MF, Rosano G, Seferovic P, Stromberg A. Self-care of heart failure patients: practical management recommendations from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2021 Jan;23(1):157-174. doi: 10.1002/ejhf.2008. Epub 2020 Oct 20. PMID 32945600
- [Result] Rahmani A, Vahedian-Azimi A, Sirati-Nir M, Norouzadeh R, Rozdar H, Sahebkar A. The Effect of the Teach-Back Method on Knowledge, Performance, Readmission, and Quality of Life in Heart Failure Patients. Cardiol Res Pract. 2020 Nov 23;2020:8897881. doi: 10.1155/2020/8897881. eCollection 2020. PMID 33299604
- [Result] Ho CC, Clochesy JM, Madigan E, Liu CC. Psychometric evaluation of the Chinese version of the Minnesota Living with Heart Failure Questionnaire. Nurs Res. 2007 Nov-Dec;56(6):441-8. doi: 10.1097/01.NNR.0000299849.21935.c4. PMID 18004191
- [Result] Wong EL, Cheung AW, Wong AY, Xu RH, Ramos-Goni JM, Rivero-Arias O. Normative Profile of Health-Related Quality of Life for Hong Kong General Population Using Preference-Based Instrument EQ-5D-5L. Value Health. 2019 Aug;22(8):916-924. doi: 10.1016/j.jval.2019.02.014. Epub 2019 Jul 27. PMID 31426933
- [Result] Sebern MD. Refinement of the Shared Care Instrument-Revised: a measure of a family care interaction. J Nurs Meas. 2008;16(1):43-60. doi: 10.1891/1061-3749.16.1.43. PMID 18578109
- [Result] Chen S, Zheng S, Wang X, Zhang X, Fa T, Fu L, Zang X, Zhao Y. Linguistic and Psychometric Validation of the Chinese Version of the Control Attitudes Scale-Revised in Patients With Chronic Heart Failure. J Cardiovasc Nurs. 2021 Jul-Aug 01;36(4):349-356. doi: 10.1097/JCN.0000000000000705. PMID 32472800
- [Result] Vickerstaff V, Ambler G, King M, Nazareth I, Omar RZ. Are multiple primary outcomes analysed appropriately in randomised controlled trials? A review. Contemp Clin Trials. 2015 Nov;45(Pt A):8-12. doi: 10.1016/j.cct.2015.07.016. Epub 2015 Jul 26. PMID 26215934
- See also: Hospital Authority Statistical Report 2016-2017 — https://www3.ha.org.hk/data/HAStatistics/DownloadReport/2?isPreview=False

DOCUMENTS (1):
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT05806606/ICF_000.pdf